CLINICAL TRIAL: NCT01090843
Title: Comparison Study of IntroMedic®'s MiroCam® and Olympus®' Enteropro EndoCapsule®
Brief Title: Video Capsule Endoscopy (VCE) Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Dolak, MD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: EK 961/2009
Record Dates: First submitted 2010-03-22; First posted 2010-03-23 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Bleeding; Anemia; Diarrhea
Keywords: Obscure digestive bleeding (ODB); Chronic anaemia of unknown origin; Chronic diarrhoea
MeSH Terms: conditions — Hemorrhage; Anemia; Diarrhea | interventions — Videotape Recording; Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Video capsule endoscopy (VCE) — In the context of video capsule endoscopy the patient will swallow the first capsule after successful mounting of adhesive electrodes and registering tool of both capsule products. The second capsule will be swallowed two hours later. The two capsules used in our investigation are the MiroCam® (product of IntroMedic®, Seoul, Korea) and the Enteropro EndoCapsule® (product of Olympus®, Tokyo, Japan). To reduce bias made up by the sequence of the capsules used, we will randomize the capsule positions at each examination, following a computer generated list.
Device: MiroCam — In the context of video capsule endoscopy the patient will swallow the first capsule after successful mounting of adhesive electrodes and registering tool of both capsule products. The second capsule will be swallowed two hours later. The two capsules used in our investigation are the MiroCam® (product of IntroMedic®, Seoul, Korea) and the Enteropro EndoCapsule® (product of Olympus®, Tokyo, Japan). To reduce bias made up by the sequence of the capsules used, we will randomize the capsule positions at each examination, following a computer generated list.
Device: Enteropro EndoCapsule — In the context of video capsule endoscopy the patient will swallow the first capsule after successful mounting of adhesive electrodes and registering tool of both capsule products. The second capsule will be swallowed two hours later. The two capsules used in our investigation are the MiroCam® (product of IntroMedic®, Seoul, Korea) and the Enteropro EndoCapsule® (product of Olympus®, Tokyo, Japan). To reduce bias made up by the sequence of the capsules used, we will randomize the capsule positions at each examination, following a computer generated list.

SUMMARY:
MiroCam® is the new video capsule endoscope of IntroMedic®. By using a novel transmission technology it promises a longer battery life expectancy with consequential impact on the length of the video recorded for diagnostic evaluation. As the investigators know about the shortcoming of battery life expectancy from many capsule examinations that were inconclusive because the ileocaecal transit was not filmed, the investigators would appreciate to have a capsule with extended video recording to improve the diagnostic yield of capsule examinations. Therefore the investigators want to compare MiroCam® to our routinely used Olympus® Enteropro EndoCapsule® in the context of a half-year clinical trial. Focussing on the total video length as well as on the rate of video-recorded ileocaecal transitions as surrogate parameters the investigators want to find out whether one of the two products provides superior diagnostic information in order to reduce the amount of inconclusive examinations.

DETAILED DESCRIPTION:
Introduction

Video capsule endoscopy (VCE) is an important tool in the diagnostic management of several gastrointestinal (GI) disorders. Taking a video while passing the GI tract, VCE is the only technique providing image information of the whole small bowel. It is a comfortable and safe procedure; complications due to capsule retention are rare [1]. The main disadvantage of VCE is made up by its only dependence on macroscopic information. Therefore it can not be reliably used for the detection of disorders that need histological confirmation. However, lots of macroscopic pathologies can be diagnosed or excluded by VCE. Above all, obscure digestive bleeding (ODB) has become the main indication for the use of VCE [2].

Independent from the type of bowel preparation used, the ileocaecal transit cannot be visualized in up to 20 percent of VCE examinations, which means the loss of diagnostic information of the last intestinal parts [3]. Risk factors of such incomplete VCE include previous small-bowel surgery, hospitalization, moderate or poor bowel cleansing and a gastric transit time longer than 45 minutes [4]. Especially in the latter case, the success of the examination is determined by the battery life expectancy of the capsule technology used [5].

The new MiroCam®, a brand of IntroMedic®, is advertised to have a longer battery life expectancy than competitive products throughout the market. To prove this pronouncement, a pilot-study of 16 patients was presented by He Man Kim at the UEGW 2008, comparing MiroCam® to Given®'s PillCam® by sequential application of both capsules. Although the battery life expectancy of MiroCam® was significantly higher, there was no significant difference in the diagnostic yield of both products [6]. Currently a similar comparison study between MiroCam® and Pill Cam® is ongoing in France, involving a higher amount of patients [unpublished data].

Study Aims

In this prospective study we want to compare IntroMedic®'s MiroCam® to Olympus® Enteropro EndoCapsule® which was so far routinely used at our department. We want to investigate whether one of the two products provides superior diagnostic information about the small bowel. The primary endpoint will be the total video length registered as well as the rate of successful ileocoecal transitions during ongoing video registration. The secondary end point will be the number of pathologies detected by each capsule. If there will be a significant difference between the two tested products, preferred usage of the superior product may improve the diagnostic yield of future examinations by avoiding incomplete video registration of the small bowel.

Study Design

Prospective Study without randomisation or blinding

Study Population

Patients transferred to our unit to undergo video capsule endoscopy because of

* Obscure digestive bleeding (ODB)
* Chronic anaemia of unknown origin
* Chronic diarrhoea

Exclusion criteria:

* Patients age below 18 years
* Patients presenting with contraindications to video capsule endoscopy which are already known gastrointestinal stenoses, already known gastrointestinal adhesions, already known diverticula of the small bowel, already known severe or diabetes induced intestinal hypomotility
* Refusal to participate in the study

Methods

Our investigation will be performed at the Medical University of Vienna, department of medicine III, clinical division of gastroenterology and hepatology. Patient recruitment will start on the 1st of January 2010. The study will last for six month. The number of patients included within this period will be around 50, based on the current amount of VCE examinations performed at our department.

All patients who fulfil the listed inclusion criteria, will receive the patient information form of this study together with the routine informed consent form of VCE. Potentially occurring questions about the course of the examination, data acquisition and processing in context of the study will be answered by medical professionals.

As routine preparation for VCE, patients will receive 2 litres of washout solution on the previous day of their examination. At the day of the procedure fasting is required. The patient will swallow the first capsule after successful mounting of adhesive electrodes and registering tool of both capsule products. The second capsule will be swallowed two hours later - to our knowledge the first capsule will have already passed the gastro-duodenal transit at this time. The two capsules used in our investigation are the already mentioned MiroCam® (product of IntroMedic®, Seoul, Korea) and the Enteropro EndoCapsule® (product of Olympus®, Tokyo, Japan). To reduce bias made up by the sequence of the capsules used, we will randomize the capsule positions at each examination, following a computer generated list. After both capsules have been swallowed, fasting has to be continued for four hours to prevent image interference of VCE.

Risk/Benefit Assessment

The safety of both products used within our investigation was already proved in former clinical trials [7, 8]. For the patients enrolled in our study the potentially higher risk of complications will be made up for the expected increase of diagnostic yield that will be implicated by the evaluation of two different bowel videos. The only notable discomfort for patients participating in our investigation will be caused by the rather high amount of adhesive electrodes necessary for both capsules. There should not be any interference of the two video signals as already shown in former investigations [6,9].

ELIGIBILITY:
Inclusion Criteria:

Patients transferred to our unit to undergo video capsule endoscopy because of

* Obscure digestive bleeding (ODB)
* Chronic anaemia of unknown origin
* Chronic diarrhoea

Exclusion Criteria:

* Patients age below 18 years
* Patients presenting with contraindications to video capsule endoscopy which are already known gastrointestinal stenoses, already known gastrointestinal adhesions, already known diverticula of the small bowel, already known severe or diabetes induced intestinal hypomotility
* Refusal to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Total video length | 6 months
  The primary endpoint will be the total video length registered as well as the rate of successful ileocoecal transitions during ongoing video registration.

SECONDARY OUTCOMES:
Diagnostic yield | 6 months
  The secondary end point will be the number of pathologies detected by each capsule.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Puespoek, MD, Study Director — Medical University of Vienna; Werner Dolak, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Medicine III., Clinical Division of Gastroenterology and Hepatology, Vienna, Austria

REFERENCES:
- [Background] Munoz-Navas M. Capsule endoscopy. World J Gastroenterol. 2009 Apr 7;15(13):1584-6. doi: 10.3748/wjg.15.1584. PMID 19340899
- [Background] Nakamura T, Terano A. Capsule endoscopy: past, present, and future. J Gastroenterol. 2008;43(2):93-9. doi: 10.1007/s00535-007-2153-6. Epub 2008 Feb 29. PMID 18306982
- [Background] Kalantzis C, Triantafyllou K, Papadopoulos AA, Alexandrakis G, Rokkas T, Kalantzis N, Ladas SD. Effect of three bowel preparations on video-capsule endoscopy gastric and small-bowel transit time and completeness of the examination. Scand J Gastroenterol. 2007 Sep;42(9):1120-6. doi: 10.1080/00365520701251601. PMID 17710680
- [Background] Westerhof J, Weersma RK, Koornstra JJ. Risk factors for incomplete small-bowel capsule endoscopy. Gastrointest Endosc. 2009 Jan;69(1):74-80. doi: 10.1016/j.gie.2008.04.034. Epub 2008 Aug 8. PMID 18691709
- [Background] Sanchez-Yague A. Risk factors for incomplete small-bowel capsule endoscopy: should capsule retention be considered independently? Gastrointest Endosc. 2009 Oct;70(4):820; author reply 820. doi: 10.1016/j.gie.2009.02.018. No abstract available. PMID 19788996
- [Background] He Man Kim. Sequential capsule endoscopy of two different capsule endoscopes, MiroCam and Pillcam SB1, without interference: a pilot study. UEGW Oct 21, 2008.
- [Background] Bang S, Park JY, Jeong S, Kim YH, Shim HB, Kim TS, Lee DH, Song SY. First clinical trial of the "MiRo" capsule endoscope by using a novel transmission technology: electric-field propagation. Gastrointest Endosc. 2009 Feb;69(2):253-9. doi: 10.1016/j.gie.2008.04.033. Epub 2008 Jul 21. PMID 18640676
- [Background] Gheorghe C, Iacob R, Bancila I. Olympus capsule endoscopy for small bowel examination. J Gastrointestin Liver Dis. 2007 Sep;16(3):309-13. PMID 17925927
- [Background] Cave DR, Fleischer DE, Leighton JA, Faigel DO, Heigh RI, Sharma VK, Gostout CJ, Rajan E, Mergener K, Foley A, Lee M, Bhattacharya K. A multicenter randomized comparison of the Endocapsule and the Pillcam SB. Gastrointest Endosc. 2008 Sep;68(3):487-94. doi: 10.1016/j.gie.2007.12.037. Epub 2008 Apr 14. PMID 18410941